CLINICAL TRIAL: NCT04951700
Title: Aging and Disease Course: Contributions to Lifespan Neurobiology of Schizophrenia
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elena Ivleva, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-0413; R01MH127317 (NIH)
Record Dates: First submitted 2021-06-01; First posted 2021-07-07 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Aging; Disease Course; Biomarker; Neuroimaging; Cognitive Dysfunction
MeSH Terms: conditions — Schizophrenia; Disease Progression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Schizophrenia: Women and men, all races and ethnicities, aged 18-65 years, meeting diagnostic DSM-5 criteria for schizophrenia or schizoaffective disorder.
  Interventions: Other: Other
- Healthy Controls: Women and men, all races and ethnicities, aged 18-75 years, without personal history of lifetime psychiatric disorders, or a family history of psychotic disorders in 1st- or 2nd-degree relatives.
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — This is not an intervention study

SUMMARY:
The 2020 NIMH Strategic Plan for Research calls for investigations targeting neurobiology of mental illness across the lifespan. Growing evidence suggests that lifespan neurobiology of schizophrenia (SZ) incorporates two distinct dimensions: aging and disease course. However, their clinical correlates, associated biomarker trajectories, and implications for treatment are unknown. This study will investigate differential aspects of SZ neurobiology captured by aging and disease course, in order to develop specific biomarkers which may offer actionable targets for SZ stage-dependent intervention. The study is predicated on a novel mechanistic Model of SZ Trajectories across the Adult Lifespan, positing distinct biological fingerprints within the anterior limbic system for aging and disease course in SZ: (1) alterations in the circuit's function and structure that occur earlier in the lifespan and are larger in magnitude than the alterations expected with normal aging (accelerated aging dimension); and (2) regionally-specific anterior limbic "hyperactivity" in early SZ, with a subsequent transformation into "hypoactivity" in advanced SZ (disease course dimension). In a sample of SZ and matched healthy controls (n=168, 84/group) aged 18-75 years the investigators will ascertain a broad panel of biomarkers [via multimodal brain imaging: optimized 1H-MRS, high-resolution task-based fMRI, perfusion (Vascular Space Occupancy) and structural MRI], along with comprehensive cognitive and clinical assessments. All measures will be acquired at baseline and repeated at 2-year longitudinal follow-up. Using cutting-edge computational approaches, the study will examine (i) effects of aging and SZ course on anterior limbic system biomarkers; (ii) lifespan trajectories for different biomarkers; (iii) patterns of limbic system biomarkers in age- and SZ course-based subgroups (e.g., Younger vs. Older, Early-Course vs. Advanced SZ), as well as in data-driven subgroups (e.g., those with vs. without accelerated aging profiles); and (iv) associations between biomarkers and cognitive and clinical outcomes. This research will advance the field by providing novel biomarkers that capture unique neurobiological contributions of aging and disease course in SZ, and will motivate future studies on SZ mechanisms across the lifespan and development of precision treatments.

DETAILED DESCRIPTION:
Specific Aims: In order to investigate aging and disease course dimensions in SZ, the study will ascertain a broad panel of biomarkers using multimodal brain imaging, along with comprehensive cognitive and clinical measures, which will allow integration of in vivo molecular; circuit structure and function; and clinical levels of system pathology.

Aim 1. In vivo Molecular Biomarkers. Examine age- and disease course-dependent effects on excitatory and inhibitory 1H-MRS-based biomarkers in the anterior limbic system in SZ. SZ and CON (n=84/group) will undergo novel triple-refocusing 1H-MRS with Glutamate (Glu), GABA and broader metabolite measures from bilateral Hipp and mPFC. Hypothesis 1.1: SZ will show declines in Hipp-mPFC Glu and GABA along the lifespan, with significantly earlier and larger reductions than those observed in CON. Hypothesis 1.2: SZ will show distinct Hipp-mPFC Glu and GABA markers along the disease course, with significantly elevated or equivalent Glu, and reduced GABA levels, in early SZ, and reduced Glu and GABA in advanced SZ, compared to CON.

Aim 2. Functional Circuit Biomarkers. Examine age- and disease course-dependent effects on intrinsic and task-based activation biomarkers in the anterior limbic circuit in SZ, using high resolution perfusion [Vascular Space Occupancy] and functional MRI with an episodic memory [Pattern Separation] task, respectively. Hypothesis 2.1: SZ will show declines in Hipp-mPFC intrinsic and task-based activity along the lifespan, with significantly earlier and larger reductions than those in CON. Hypothesis 2.2: SZ will show distinct Hipp-mPFC intrinsic and task-dependent activity signatures across the disease course, with significantly elevated or equivalent regional activation in early SZ, and reduced activation in advanced SZ, compared to CON.

Aim 3. Structural Circuit Biomarkers. Examine age- and disease course-dependent effects on structural biomarkers in the anterior limbic system in SZ, using high resolution structural MRI. Hypothesis 3.1: SZ will show declines in cortical thickness and volume in Hipp, mPFC and broader fronto-temporal regions across the lifespan, with significantly earlier and larger reductions than those in CON. Hypothesis 3.2: SZ will show distinct fronto-temporal alterations along the disease course, with modestly reduced cortical thickness and volume measures in early SZ and larger reductions in advanced SZ, compared to CON.

The investigators also predict that molecular, functional, and structural alterations in the anterior limbic system will be associated with impaired episodic memory and broader cognitive dysfunction in SZ, with declining cognition along both the lifespan and SZ course.

This research will advance the field by providing novel biomarkers that capture unique neurobiological contributions of aging and disease course in SZ, and will motivate future studies on SZ mechanisms across the lifespan, and the development of relevant precision treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age (SZ); 18-75 years of age (CON)
* Women and men
* All races and ethnicities
* Psychiatric diagnoses:

Patient participants (SZ): Meet DSM-5 criteria for schizophrenia or schizoaffective disorder Healthy control participants (CON): No personal history of lifetime psychiatric disorders, or a family history of psychotic disorders in 1st-or 2nd- degree relatives

* Able to read, speak, and understand English
* Able and willing to provide written informed consent; and willing to commit to the study protocol, including 2-year longitudinal follow-up

Exclusion Criteria:

• Compromised cognitive function: Both SZ and CON participants: Estimated premorbid intellectual ability <75 age-corrected score on Wide Range Achievement Test-4/Word Reading Subtest (WRAT-4) CON participants: <26 score on the Montreal Cognitive Assessment (MoCA)

* Neurological or medical disorder that may affect brain function (history of stroke, head injury with a loss of consciousness >10 min, seizure disorder, AIDS, poorly controlled hypertension, poorly controlled diabetes, decompensated lung disease, etc.)
* Co-morbid DSM-5 diagnosis of drug/alcohol use disorder in prior 3 months
* Current treatment with benzodiazepine or non-benzodiazepine sedatives/hypnotics, and/or anticonvulsants
* Presence of ferromagnetic objects in body
* Weight or body size exceeding MRI scanner capacity [>300 lbs]
* Claustrophobia in MRI scanner
* Pregnant women
* Breastfeeding women (VASO scan will not be administered. All other imaging modalities are safe to administer.)
* Impaired kidney function: Glomerular Filtration Rate (GFR) < 30 ml/min/1.73m2 (VASO scan will not be administered due to an association between Gadolinium-based MR contrast use and Nephrogenic Systemic Fibrosis in individuals with severely impaired renal function. All other imaging modalities are safe to administer.)
* History of hypersensitivity to any MRI contrast agent (VASO scan will not be administered. All other imaging modalities are safe to administer.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include individuals with psychotic disorders (schizophrenia or schizoaffective disorder) and healthy comparison participants (individuals without personal history of lifetime psychiatric disorders, or a family history of psychotic disorders in 1st- or 2nd-degree relatives). Participants will be women and men, all races and ethnicities. Participants with schizophrenia/schizoaffective disorder will be aged 18-65 years, healthy comparison participants will be aged 18-75 years.
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Effects of aging and disease course on excitatory and inhibitory biomarkers in the anterior limbic system in schizophrenia (SZ) and healthy controls (CON) (Aim1 Outcomes). | 2 years
  SZ and CON (n=84/group) will undergo novel triple-refocusing Magnetic Resonance Spectroscopy (1H-MRS) with Glutamate, GABA and broader metabolite measures from the anterior limbic system structures (bilateral hippocampi (Hipp) and medial prefrontal cortex (mPFC)), at baseline and 2-year longitudinal follow-up. Hypothesis 1.1: SZ will show declines in Glutamate and GABA in the Hipp and mPFC along the lifespan, with significantly earlier and larger reductions than those observed in CON. Hypothesis 1.2: SZ will show distinct Hipp-mPFC Glutamate and GABA markers along the disease course, with significantly elevated or equivalent Glutamate, and reduced GABA levels, in early SZ, and reduced Glutamate and GABA in advanced SZ, compared to CON.
Effects of aging and disease course on intrinsic activity biomarkers [VASO-based Cerebral Blood Volume (CBV)] in the anterior limbic circuit in SZ and CON (Aim2 Outcome). | 2 years
  SZ and CON will undergo high-resolution brain perfusion imaging (VASO) at baseline and 2-year longitudinal follow-up. Hypothesis 2.1: SZ will show declines in Hipp-mPFC CBV along the lifespan, with significantly earlier and larger reductions than those observed in CON. Hypothesis 2.2: SZ will show distinct Hipp-mPFC CBV signatures across the disease course, with significantly elevated or equivalent CBV in early SZ, and reduced CBV in advanced SZ, compared to CON.
Effects of aging and disease course on memory task-driven activation biomarkers [fMRI with Pattern Separation task] in the anterior limbic circuit in SZ and CON (Aim2 Outcome). | 2 years
  SZ and CON will undergo high-resolution brain fMRI with associational memory (Pattern Separation) task at baseline and 2-year longitudinal follow-up. Hypothesis 2.1: SZ will show declines in regional activation (BOLD signal) with Lure>Repetition contrast along the lifespan, with significantly earlier and larger reductions than those in CON. Hypothesis 2.2: Within the disease course dimension, early SZ will show increased activation with a loss of activation modulation (e.g., increased BOLD signal with both Lures and Repetitions), with a subsequent decline in activation in mid-course and advanced SZ, compared to CON. We predict that these activation effects will be preset in the Hipp DG/CA3 and in a broader circuit supporting pattern separation operations (i.e., mPFC, parahippocampal, retrosplenial cortex).
Effects of aging and disease course on cortical thickness biomarkers in the anterior limbic system in SZ and CON (Aim3 Outcomes). | 2 years
  SZ and CON will undergo high-resolution structural brain MRI, at baseline and 2-year longitudinal follow-up. Hypothesis 3.1: SZ will show declines in FreeSurfer-based cortical thickness in Hipp, mPFC and broader fronto-temporal regions across the lifespan, with significantly earlier and larger reductions than those in CON. Hypothesis 3.2: SZ will show distinct fronto-temporal alterations along the disease course, with modestly reduced cortical thickness in early SZ and larger reductions in advanced SZ, compared to CON.
Effects of aging and disease course on gray matter volume biomarkers in the anterior limbic system in SZ and CON (Aim3 Outcomes). | 2 years
  SZ and CON will undergo high-resolution structural brain MRI, at baseline and 2-year longitudinal follow-up. Hypothesis 3.1: SZ will show declines in gray matter volumes (measured with FreeSurfer and Voxel-Based Morphometry) in Hipp, mPFC and broader fronto-temporal regions across the lifespan, with significantly earlier and larger reductions than those in CON. Hypothesis 3.2: SZ will show distinct fronto-temporal alterations along the disease course, with modestly reduced gray matter volume in early SZ and larger reductions in advanced SZ, compared to CON.

OTHER OUTCOMES:
Associations between brain MRI and cognitive and clinical measures. | 2 years
  A broad panel of cognitive (Wide Range Achievement Test/Reading Subtest (WRAT-4/Reading Subtest), Brief Assessment of Cognition in Schizophrenia (BACS), California Verbal Learning Test-2nd Edition (CVLT-II), Ruff-Light Trial Learning Test (RULIT)) and clinical (socio-demographic information, psychiatric, medical and treatment history, family history, concomitant medications, Structured Clinical Interview for DSM-5 (SCID-5), Global Assessment of Functioning (GAF), Birchwood Social Functioning Scale (SFS), Positive and Negative Syndrome Scale PANSS), Lifetime Dimensions of Psychosis Scale (LDPS), Ciompi's Observed Course Chart, Fagerstrom Test for Nicotine Dependence) assessments will be collected from SZ and CON, at baseline and 2-year longitudinal follow-up. Associations between multimodal brain MRI measures and cognitive and clinical measures will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Elena I. Ivleva, MD, PhD, Principal Investigator — UT Southwestern Medical Center, Department of Psychiatry
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States